CLINICAL TRIAL: NCT05441306
Title: Personal Health Libraries for Formerly Incarcerated Individuals
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Library of Medicine (NLM) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2000028862; 1R01LM013477-01 (NIH)
Record Dates: First submitted 2022-06-28; First posted 2022-07-01 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Personal Health Information; Incarcerated Individuals

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Access to Personal Health Library (PerHL) + MyChart (Experimental): Participants randomized to the PerHL arm will have access to PerHL and the standard of care patient portal (Epic®MyChart).
  Interventions: Device: Personal Health Library (PerHL) + MyChart
- Control - MyChart (Active Comparator): Participants randomized to the control arm will receive the standard of care patient portal (Epic®MyChart).
  Interventions: Device: Epic®MyChart

INTERVENTIONS:
Device: Personal Health Library (PerHL) + MyChart — Participants randomized to the PerHL arm will have access to PerHL + the standard of care patient portal (Epic®MyChart).
  Arms: Access to Personal Health Library (PerHL) + MyChart
Device: Epic®MyChart — Participants randomized to the control arm will receive the standard of care patient portal (Epic®MyChart).
  Arms: Control - MyChart

SUMMARY:
This is a randomized pilot study to test the acceptance and use of PerHL among formerly incarcerated individuals

DETAILED DESCRIPTION:
Eligible participants will be enrolled after providing informed consent .Participants will then complete a baseline assessment. After the interview, eligible participants will be randomly assigned to the intervention or control group. The research assistant (RA) will be blinded to the randomization allocation until after the consent process. For the purposes of this study, permuted block randomization with random block sizes of 2, 4 and 6 will be used.

Intervention: Those randomized to the intervention arm will have access to PerHL. The intervention group will watch a demonstration by the RA and will practice using PerHL for 10-15 minutes, i.e. taking a picture of a document and uploading to PerHL, entering specific information, voice recording an appointment reminder. The RA will be responsible for providing technical support and assist with the need for initial support, e.g. phone-call or text-based support. At baseline, participants will be asked to provide a list of every organization they visited that may have health and health-related social information on them and receive consent to request their information to be sent to the participant and the study team on their behalf.

Control: Participants randomized to the control arm will receive the standard of care patient portal (Epic®MyChart). The RA will give them an informational pamphlet outlining key features of the patient portal and guide them through the steps for signing up for a MyChart account, assist them to sign up, add the standard patient portal MyChart app to their phone, and provide them with the MyChart technical support hotline.

Study Procedures: During the intervention phase, all participants will meet with the RA at baseline, 1- and 3 months. During the study, each participant will be asked to provide at least 5 verified locators who are likely to have knowledge of their whereabouts throughout follow-up. Each participant will be provided with $50 payment to participants for each completion of surveys at baseline, 1, 3 months. In addition, participants will be given $10 each month to travel to a location with free wireless so their information can be uploaded to the cloud and a list of available locations. In total, each participant will receive $180 for participation.

For the 1- and 3-month follow-up period, the RA will ask participants to bring information collected and uploaded in PerHL and additional information that is important to the participant but was not uploaded.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* English-speaking
* have at least one chronic condition
* engaged in primary care in the community
* have been released from a correctional facility in the past year.

Exclusion Criteria:

* visual impairments
* cognitive impairments
* language barriers
* planned relocation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Acceptance - Intention to use | 1 month post enrollment
  Assess intention to use the app developed for the project. Intention to use will be assessed by a survey conducted in person. This survey item is in development.
Acceptance - Intention to use | 3 month post enrollment
  Assess intention to use the app developed for the project. Intention to use will be assessed by a survey conducted in person. This survey item is in development.
Use of Personal health information technology | 1 month post enrollment
  Assess the number of times the personal health information app was accessed each week and the duration of time on the system per week. This will be assessed using tracking functionality built into the app.
Use of Personal health information technology | 3 month post enrollment
  Assess the number of times the personal health information app was accessed each week and the duration of time on the system per week. This will be assessed using tracking functionality built into the app.

SECONDARY OUTCOMES:
Perceived ease of use for the app | 1 month post enrollment
  Assess how easy it was for the participant to use the app. Perceived ease of use will be assessed by self-report survey. This survey item is in development.
Perceived ease of use for the app | 3 month post enrollment
  Assess how easy it was for the participant to use the app. Perceived ease of use will be assessed by self-report survey. This survey item is in development.
Perceived usefulness of the app | 1 month post enrollment
  Assess how useful the participant found app to be. Perceived usefulness will be assessed by self-report survey. This survey item is in development.
Perceived usefulness of the app | 3 month post enrollment
  Assess how useful the participant found app to be. Perceived usefulness will be assessed by self-report survey. This survey item is in development.
Attitude towards use of technology | 1 month post enrollment
  Assess the participant's attitude towards using technology. Attitude towards technology will be assessed by self-report survey. This survey item is in development.
Attitude towards use of technology | 3 month post enrollment
  Assess the participant's attitude towards using technology. Attitude towards technology will be assessed by self-report survey. This survey item is in development.
Completeness of data | 1 month post enrollment
  Assess the proportion of health system data sources received by study team and/or patient (#organizational data received/ #organizational requests made), assess type of data received (# of medication list received/ requested or # of allergies received/requests made) to determine completeness of data.
Completeness of data | 3 month post enrollment
  Assess the proportion of health system data sources received by study team and/or patient (#organizational data received/ #organizational requests made), assess type of data received (# of medication list received/ requested or # of allergies received/requests made) to determine completeness of data.
General self-efficacy | 1 month post enrollment
  Assess participant self-efficacy. Self-efficacy will be assessed by self-report survey. This survey item is in development.
General self-efficacy | 3 month post enrollment
  Assess participant self-efficacy. Self-efficacy will be assessed by self-report survey. This survey item is in development.
Medication adherence | 1 month post enrollment
  Medication Adherence will be measured by personal health information technology use (MyChart) at Yale New Haven Hospital, medication adherence (as measured by ninety-day medication refill).
Medication adherence | 3 month post enrollment
  Medication Adherence will be measured by personal health information technology use (MyChart) at Yale New Haven Hospital, medication adherence (as measured by ninety-day medication refill).
Engagement in primary care | 1 month post enrollment
  Engagement in primary care will be measured by personal health information technology use (MyChart) at Yale New Haven Hospital, engagement in primary care (as measured by appointments made) via MyChart systems.
Engagement in primary care | 3 month post enrollment
  Engagement in primary care will be measured by personal health information technology use (MyChart) at Yale New Haven Hospital, engagement in primary care (as measured by appointments made) via MyChart systems.

CONTACTS AND LOCATIONS:
Overall Officials: Karen Wang, MD, MHS, Principal Investigator — Yale University
Locations (1):
- Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No